CLINICAL TRIAL: NCT01945346
Title: A Double-Blind, Randomised, Exploratory Study to Investigate the Safety, Efficacy and Pharmacokinetics of PRX167700 in Subjects With Knee Osteoarthritis.
Brief Title: An Exploratory Study of PRX167700 in Patients With Knee Osteoarthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Proximagen Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 167700-002CL
Record Dates: First submitted 2013-09-13; First posted 2013-09-18 (Estimated); Last update posted 2015-08-26 (Estimated); Status verified 2015-08

CONDITIONS: Osteoarthritis, Knee
Keywords: PRX167700; Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- PRX167700 (Experimental)
  Interventions: Drug: PRX167700
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PRX167700 — Oral capsule
  Arms: PRX167700
Drug: Placebo — Oral capsule
  Arms: Placebo

SUMMARY:
This is an exploratory study to evaluate a new anti-inflammatory drug, PRX167700, in subjects with painful osteoarthritis of the knee.

The purpose of this study is to investigate if PRX167700 improves the pain from osteoarthritis of the knee, and to assess its safety and tolerability. The study will also investigate PRX167700 pharmacokinetics.

DETAILED DESCRIPTION:
Up to 74 subjects will receive either PRX167700 or placebo (a dummy treatment) for 15 days. Subjects will need to stop taking their usual pain reliever medicines for at least 7 days before starting treatment to induce a 'flare' in osteoarthritis symptoms (but they will be allowed to continue to use paracetamol for immediate pain relief as needed throughout the trial). The effect of PRX167700 or placebo on knee pain will be assessed before and after exercise on Days 1, 3, 7 and 14. On Day 15, blood samples will be collected to measure levels of PRX167700 and assess its activity.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) between 20 and 35 kg/m2, inclusive.
* Symptomatic primary OA of the knee for at least 3 months prior to Screening according to the American College of Rheumatology (ACR) criteria.
* Diagnosis of OA of the knee based on ACR criteria with X-ray confirmation (a Kellgren-Lawrence X-ray grade of ≥2) in the target knee joint.
* Use of analgesics for the treatment of knee OA for at least 4 out of 7 days in each of the 4 weeks preceding the Screening visit.
* Willing and able to discontinue all current analgesic therapy, including over the counter (OTC) pain medications and topical analgesics for OA pain, for a period beginning at Screening and continuing for the entire duration of the study.
* Able to walk 100 metres on a flat course without rest and unaided.
* A self-rated Pain Intensity score in the target knee joint of between 3 and 8, inclusive, immediately after a timed 100 metres walk on a flat course.
* Able to provide written informed consent to participate in the study and, in the opinion of the investigator, able to read, comprehend and record information as required by the protocol.

Exclusion Criteria:

* Secondary causes of arthritis of the knee, disease of the spine or of lower extremity joints (other than OA), knee pain characteristic of neuropathic pain.
* Lower extremity surgery (including arthroscopy) within 6 months prior to Screening or scheduled for surgery of any kind during the study.
* Significant injury to the target knee joint within 12 months prior to Screening.
* Known history of hypersensitivity or intolerance to paracetamol or lactose.
* Oral corticosteroids within 1 month of Screening
* Therapeutic injections into the target knee joint within previous 3 months. Intra-articular corticosteroid injections into any other site within 1 month or intra-muscular corticosteroid injections within 3 months.
* Start or change in dosing regimen of other therapies for OA within 3 months of Screening.
* Start or change in an established physiotherapy programme within 2 weeks of Screening (Visit 1) or during the course of the study. An established physiotherapy program may be continued throughout the study period if unchanged in frequency and intensity.
* Any significant clinical or biological abnormality (other than those related to OA) which would preclude safe participation in this study.

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2013-09; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Pain Intensity | Study Days 0 [Baseline], 1, 3, 7 and 14
  Measured at rest and after exercise at 1, 2 and 3 hours post-dose. Measured using 11-point numerical rating scale (NRS)ranging from 0 to 10 where 0 represents no pain and 10 represents the worst possible pain

SECONDARY OUTCOMES:
Efficacy: | Study Days 0 [Baseline], 1, 3, 7 and 14
  * Western Ontario and McMaster Universities (WOMAC)Questionnaire total score and subscales;
  * Patient Global Impression of Change;
  * Time to complete exercise;
  * Serum C-reactive protein levels;
  * Rescue medication use.
Safety | 15 days
  Safety and tolerability will be evaluated by assessing adverse events (AEs), clinical laboratory data, physical examinations, vital signs, and electrocardiograms (ECGs).

OTHER OUTCOMES:
Pharmacokinetics | Day 15
  Plasma concentration-time profiles and pharmacokinetic parameters, including (but not limited to) Cmax, tmax, area under the plasma concentration vs. time curve from time zero over the dosing interval, area under the concentration-time curve over the dose interval and to infinity, and, if possible, t½.will be determined.
Pharmacodynamics | Day 15
  Biomarker activity following dosing

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Proximagen Limited
Locations (5):
- United Kingdom (5):
  - Proximagen Investigational Site, Birmingham
  - Proximagen Investigational Site, Lancashire
  - Proximagen Investigational Site, Liverpool
  - Proximagen Investigational Site, Manchester
  - Proximagen Investigational Site, Reading